CLINICAL TRIAL: NCT01122420
Title: Online Resources to Manage Obesity and Health Risks in an Employee Wellness Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Gretchen Purcell Jackson, MD, PhD, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100021
Record Dates: First submitted 2010-05-10; First posted 2010-05-13 (Estimated); Last update posted 2013-08-22 (Estimated); Status verified 2013-08

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Goal-Setting Tool (Experimental)
  Interventions: Other: Goal-Setting Tool
- Health Web Sites (Active Comparator)
  Interventions: Other: Health Web Sites

INTERVENTIONS:
Other: Goal-Setting Tool — Access to an online health-related goal-setting tool through the MyHealthAtVanderbilt patient portal
  Arms: Goal-Setting Tool
Other: Health Web Sites — Access to publicly available health-related web sites
  Arms: Health Web Sites

SUMMARY:
The purpose of this study is to determine whether different types of online health tools can aid overweight individuals in reducing their weight and managing their cardiovascular risk factors in the context of an employee wellness program.

ELIGIBILITY:
Inclusion Criteria:

* Vanderbilt University employee
* Completion of the 2009 Go For the Gold Health Risk Assessment (HRA)
* Obesity defined by BMI > 30
* Identification of an additional risk factor on the HRA by either (a) a personal history of diabetes, high blood pressure, or high cholesterol or (b) a reported cholesterol >= 240 mg/dl, blood glucose >= 126 mg/dl, a systolic blood pressure >= 140 mm Hg, or a diastolic blood pressure >= 90 mm Hg
* Permission to be contacted regarding health on the HRA

Exclusion Criteria:

* Pregnant females and those who become pregnant prior to completion of the study
* Age younger than 18 years or older than 65 years
* Non English speaking individuals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in body mass index | At enrollment and at 6 months
Change in excess body weight | At enrollment and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen P Jackson, M.D., Ph.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States